CLINICAL TRIAL: NCT01189500
Title: An Open-Label, 2-Period Sequential Drug Interaction Study To Evaluate The Effect Of A 100 Mg Dose Of Desvenlafaxine SR On The Pharmacokinetics Of Tamoxifen When Co-Administered In Healthy Post-Menopausal Female Subjects
Brief Title: Open-Label Drug Interaction Study Evaluating Desvenlafaxine Succinate Sustained Release (DVS SR) 100mg On The Pharmacokinetics Of Tamoxifen When Coadministered To Healthy Post-Menopausal Female Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B2061027; 3151A1-1206
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Pharmacokinetics
Keywords: Pharmacokinetic; safety and tolerability; genetic testing; CYP 2D6
MeSH Terms: interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tamoxifen and Desvenlafaxine SR (Experimental)
  Interventions: Drug: Tamoxifen; Drug: Tamoxifen and Desvenlafaxine Succinate Sustained Release

INTERVENTIONS:
Drug: Tamoxifen — Period 1-Tamoxifen 40mg on study day 1.
Drug: Tamoxifen and Desvenlafaxine Succinate Sustained Release — Period 2-Desvenlafaxine SR 100mg on days 1-28 with coadministration of Tamoxifen 40mg on day 7.

SUMMARY:
The goal of this study is to evaluate the effect of multiple doses of Desvenlafaxine SR on the pharmacokinetics of Tamoxifen and endoxifen when coadministered to healthy post-menopausal female subjects. This study will also evaluate the safety and tolerability of Desvenlafaxine SR and Tamoxifen when coadministered to healthy post-menopausal female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy post-menopausal female subjects, at least 45 years of age, with confirmed post-menopausal status
* Hysterectomized subjects
* Body Mass Index (BMI) less than or equal to 34.0 kg/m2
* Nonsmoker or smoker of fewer than 5 cigarettes per day as determined by history
* An informed consent document signed and dated by the subject

Exclusion Criteria:

* History of significant blood, kidney, endocrine, lung, gastrointestinal, heart, liver, psychiatric, neurologic, or allergic disease
* Presence or history of deep vein thrombosis or transient ischemic attack
* History of seizure disorder
* Presence or history of glaucoma or increased intraocular pressure
* Allergy to or unable to tolerate tamoxifen, desvenlafaxine, or venlafaxine
* History of substance abuse within 1 year of study
* A positive urine drug screen
* Treatment with an investigational drug within 30 days
* Consumption of grapefruit or grapefruit related citrus fruits
* 12 lead ECG demonstrating QTc >450 msec at screening
* Pregnant or nursing females
* Use of prescription or nonprescription drugs and dietary supplements
* History of sensitivity to heparin or heparin induced thrombocytopenia
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality
* Use of CYP 2D6 inhibitors and CYP 3A4 inhibitors/inducers

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Miami, Florida, United States

REFERENCES:
- [Derived] Nichols AI, Lubaczewski S, Liang Y, Matschke K, Braley G, Ramey T. Open-label, 2-period sequential drug interaction study to evaluate the effect of a 100-mg dose of desvenlafaxine on the pharmacokinetics of tamoxifen when coadministered in healthy postmenopausal female subjects. Int J Clin Pharmacol Ther. 2014 Oct;52(10):830-41. doi: 10.5414/CP201958. PMID 25138680

RESULTS

PARTICIPANT FLOW:
Groups:
- Tamoxifen 40 mg, Tamoxifen 40 mg + DVS SR 100 mg: Tamoxifen (TAMOX) 40 milligrams (mg) as a single oral dose Period 1 / Day 1. Desvenlafaxine sustained release (DVS SR) 100 mg as a single oral dose Period 2 / Day 1 through Day 6 (steady state) and Day 7 through Day 28. A single oral dose of Tamoxifen 40 mg coadministered with the DVS SR dose on Period 2 / Day 7.
Period: Period 1: TAMOX Alone
Arm/Group | Tamoxifen 40 mg, Tamoxifen 40 mg + DVS SR 100 mg
Started | 30
Completed | 29
Not Completed | 1
Not completed — Adverse Event | 1
Period: Period 2: Coadministration TAMOX+DVS SR
Arm/Group | Tamoxifen 40 mg, Tamoxifen 40 mg + DVS SR 100 mg
Started | 29
Completed | 28
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Tamoxifen 40 mg, Tamoxifen 40 mg + DVS SR 100 mg: Tamoxifen 40 mg as a single oral dose Period 1 / Day 1. DVS SR 100 mg as a single oral dose Period 2 / Day 1 through Day 6 (steady state) and Day 7 through Day 28. A single oral dose of Tamoxifen 40 mg coadministered with the DVS SR dose on Period 2 / Day 7.
Arm/Group | Tamoxifen 40 mg, Tamoxifen 40 mg + DVS SR 100 mg
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  45 to 64 years | 27
  ≥65 years | 3
Sex/Gender, Customized [Number; unit: participants] — Female
  participants | 30

OUTCOME MEASURES:

1. Primary Outcome: Tamoxifen Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞); measured as nanograms multiplied by hours divided by milliliters (ng*hr/mL).
Time Frame: Period 1 / Day 1: 0, 0.5, 1, 2, 3, 4, 6, 8, 12,16, 24, 48, 72, 120, 168, 216, 264, 312, 384, 456, and 528 hours after dosing; Period 2 / Day 1 and Day 7: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours; 0 hour on Day 8, 9, 10, 12, 14, 16, 18, 20, 23, 26 and 29.
Population: Pharmacokinetic (PK) parameter analysis population: all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Tamoxifen 40 mg (Period 1): Tamoxifen 40 mg as a single oral dose Period 1 / Day 1.
- Tamoxifen 40 mg + DVS SR 100 mg (Period 2): DVS SR 100 mg as a single oral daily dose Period 2 / Day 1 through Day 6 (steady state) and Day 7 through Day 28. A single oral dose of Tamoxifen 40 mg coadministered with the DVS SR dose on Period 2 / Day 7.
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 26 | 26
ng*hr/mL | 5751 (1540.1) | 5888 (1905.5)
Statistical Analysis 1: Comparison: Tamoxifen 40 mg (Period 1) vs Tamoxifen 40 mg + DVS SR 100 mg (Period 2); DVS SR 100 mg + Tamoxifen 40 mg (test) versus Tamoxifen 40 mg (reference); Test type: Superiority or Other; ratio of adjusted means = 100.69, 90% CI 2-sided [96.70 to 104.85] — Values have been back-transformed from the log scale

2. Primary Outcome: Endoxifen (Metabolite) Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) Following Endoxifen Alone and When Coadministered With DVS SR
Description: Endoxifen is a metabolite of Tamoxifen. Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 4 | 4
ng*hr/mL | 677.7 (200.42) | 505.6 (220.87)

3. Secondary Outcome: Tamoxifen Maximum Observed Concentration (Cmax) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Cmax measured as nanograms per milliliters (ng/mL).
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
ng/mL | 70.58 (16.310) | 70.33 (14.484)
Statistical Analysis 1: Comparison: Tamoxifen 40 mg (Period 1) vs Tamoxifen 40 mg + DVS SR 100 mg (Period 2); DVS SR 100 mg + Tamoxifen 40 mg (test) versus Tamoxifen 40 mg (reference); Test type: Superiority or Other; ratio of adjusted means = 99.44, 90% CI 2-sided [94.02 to 105.17] — Values have been back-transformed from the log scale

4. Secondary Outcome: Tamoxifen Time for Cmax (Tmax) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Time for maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the median.
Measure: Median (Full Range); unit: hours
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
hours | 4.00 [3.00 to 8.00] | 4.00 [3.00 to 8.00]

5. Secondary Outcome: Tamoxifen Terminal Half-life (t 1/2) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 26 | 26
hours | 250.5 (44.410) | 242.3 (51.851)

6. Secondary Outcome: Tamoxifen Apparent Clearance (CL/F) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood calculated as (Dose/AUCinf); measured as milliliters per minute (mL/min).
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: mL/min
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 26 | 26
mL/min | 115.9 (34.544) | 113.2 (44.545)

7. Secondary Outcome: Tamoxifen Apparent Volume of Distribution (Vz/F) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Calculated as Dose / (AUCinf * kel); where kel=terminal phase rate constant.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: liters
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 26 | 26
liters | 2474 (461.71) | 2321 (419.76)

8. Secondary Outcome: Endoxifen (Metabolite) Maximum Observed Concentration (Cmax) Following Tamoxifen Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
ng/mL | 1.077 (0.4528) | 1.226 (0.4956)
Statistical Analysis 1: Comparison: Tamoxifen 40 mg (Period 1) vs Tamoxifen 40 mg + DVS SR 100 mg (Period 2); DVS SR 100 mg + Tamoxifen 40 mg (test) versus Tamoxifen 40 mg (reference); Test type: Superiority or Other; ratio of adjusted means = 92.04, 90% CI 2-sided [84.71 to 100.00] — Values have been back-transformed from the log scale

9. Secondary Outcome: Endoxifen (Metabolite) Time for Cmax (Tmax) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Time for maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the median.
Measure: Median (Full Range); unit: hours
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
hours | 216 [47.9 to 312] | 120 [47.9 to 384]

10. Secondary Outcome: Endoxifen (Metabolite) Terminal Half-life (t 1/2) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 4 | 4
hours | 207.5 (43.59) | 232.5 (56.719)

11. Secondary Outcome: Endoxifen (Metabolite) Apparent Clearance (CL/F) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: as for outcome 6
Time Frame: as for outcome 1
Population: PK parameter analysis population. Data was insufficient for analysis; not analyzable.
Measure: Geometric Mean (Standard Deviation); unit: mL/min
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Endoxifen (Metabolite) Apparent Volume of Distribution (Vz/F) Following Tamoxifen Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population. Data was insufficient for analysis; not analyzable.
Measure: Geometric Mean (Standard Deviation); unit: liters
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: N-desmethyl-tamoxifen (Metabolite) Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: N-desmethyl-tamoxifen is a metabolite of Tamoxifen. Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 4 | 7
ng*hr/mL | 8187 (1688.0) | 9329 (2236.8)

14. Secondary Outcome: N-desmethyl-tamoxifen (Metabolite) Maximum Observed Concentration (Cmax) Following Tamoxifen Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
ng/mL | 18.30 (3.7576) | 24.42 (4.3709)
Statistical Analysis 1: Comparison: Tamoxifen 40 mg (Period 1) vs Tamoxifen 40 mg + DVS SR 100 mg (Period 2); DVS SR 100 mg + Tamoxifen 40 mg (test) versus Tamoxifen 40 mg (reference); Test type: Superiority or Other; ratio of adjusted means = 112.07, 90% CI 2-sided [107.44 to 116.90] — Values have been back-transformed from the log scale

15. Secondary Outcome: N-desmethyl-tamoxifen (Metabolite) Time for Cmax (Tmax) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Time for maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the median.
Measure: Median (Full Range); unit: hours
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
hours | 35.9 [4.00 to 312] | 47.9 [4.00 to 168]

16. Secondary Outcome: N-desmethyl-tamoxifen (Metabolite) Terminal Half-life (t 1/2) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Mean (Standard Error); unit: hours
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 4 | 7
hours | 256.0 (24.042) | 265.6 (32.082)

17. Secondary Outcome: N-desmethyl-tamoxifen (Metabolite) Apparent Clearance (CL/F) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: as for outcome 6
Time Frame: as for outcome 1
Population: PK parameter analysis population. Data was insufficient for analysis; not analyzable.
Measure: Geometric Mean (Standard Deviation); unit: mL/min
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: N-desmethyl-tamoxifen (Metabolite) Apparent Volume of Distribution (Vz/F) Following Tamoxifen Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population. Data was insufficient for analysis; not analyzable.
Measure: Geometric Mean (Standard Deviation); unit: liters
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: 4-hydroxy-tamoxifen (Metabolite) Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: 4-hydroxy-tamoxifen is a metabolite of Tamoxifen. Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 25 | 26
ng*hr/mL | 117.5 (55.433) | 133.9 (62.784)
Statistical Analysis 1: Comparison: Tamoxifen 40 mg (Period 1) vs Tamoxifen 40 mg + DVS SR 100 mg (Period 2); DVS SR 100 mg + Tamoxifen 40 mg (test) versus Tamoxifen 40 mg (reference); Test type: Superiority or Other; ratio of adjusted means = 105.60, 90% CI 2-sided [99.74 to 111.81] — Values have been back-transformed from the log scale

20. Secondary Outcome: 4-hydroxy-tamoxifen (Metabolite) Maximum Observed Concentration (Cmax) Following Tamoxifen Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
ng/mL | 0.6716 (0.1649) | 0.7247 (0.1799)
Statistical Analysis 1: Comparison: Tamoxifen 40 mg (Period 1) vs Tamoxifen 40 mg + DVS SR 100 mg (Period 2); DVS SR 100 mg + Tamoxifen 40 mg (test) versus Tamoxifen 40 mg (reference); Test type: Superiority or Other; ratio of adjusted means = 108.47, 90% CI 2-sided [103.51 to 113.67] — Values have been back-transformed from the log scale

21. Secondary Outcome: 4-hydroxy-tamoxifen (Metabolite) Time for Cmax (Tmax) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Time for maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the median.
Measure: Median (Full Range); unit: hours
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
hours | 6.00 [4.00 to 12.00] | 6.00 [3.00 to 23.9]

22. Secondary Outcome: 4-hydroxy-tamoxifen (Metabolite) Terminal Half-life (t 1/2) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: PK parameter analysis population. N=number of participants contributing to the mean.
Measure: Mean (Standard Error); unit: hours
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 25 | 26
hours | 165.2 (49.699) | 177.0 (54.525)

23. Secondary Outcome: 4-hydroxy-tamoxifen (Metabolite) Apparent Clearance (CL/F) Following Tamoxifen Alone and When Coadministered With DVS SR
Description: as for outcome 6
Time Frame: as for outcome 1
Population: PK parameter analysis population. Data was insufficient for analysis; not analyzable.
Measure: Geometric Mean (Standard Deviation); unit: mL/min
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: 4-hydroxy-tamoxifen (Metabolite) Apparent Volume of Distribution (Vz/F) Following Tamoxifen Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population. Data was insufficient for analysis; not analyzable.
Measure: Geometric Mean (Standard Deviation); unit: liters
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Plasma Tamoxifen Concentration Versus Time Summary: Tamoxifen Alone and When Coadministered With DVS SR
Description: Summary statistics were to be calculated by setting concentration values below the lower limit of quantification (LLQ = 0.250 ng/mL) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) = 0.
Time Frame: Period 1 / Day 1 and Period 2 / Day 1: 0, 0.5, 1, 2, 3, 4, 6, 8, 12,16, 24, 48, 72, 120, 168, 216, 264, 312, 384, 456, and 528 hours after dosing
Population: PK concentration analysis population: all participants randomized and treated who had at least 1 concentration in at least 1 treatment period. N=number of participants contributing to the median. Period 2 / Day 1 = Day 1 of Tamoxifen dosing (Period 2 / Day 7) within the DVS SR, Tamoxifen coadministration dosing period.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
ng/mL
  0 hour | NA [NA to NA] — No observations above the lower limit of quantification. | 1.300 [0.293 to 4.66]
  0.5 hour post dose | 1.875 [0.000 to 10.3] | 4.650 [1.70 to 19.1]
  1 hour post dose | 11.45 [0.769 to 36.1] | 13.90 [3.31 to 47.8]
  2 hours post dose | 37.20 [2.55 to 74.7] | 33.60 [11.0 to 75.2]
  3 hours post dose | 54.50 [6.57 to 100] | 55.60 [17.0 to 99.4]
  4 hours post dose | 68.25 [26.9 to 95.7] | 72.20 [26.6 to 90.7]
  6 hours post dose | 58.95 [40.1 to 89.3] | 60.90 [38.5 to 90.8]
  8 hours post dose | 54.75 [32.2 to 77.8] | 56.10 [33.6 to 73.9]
  12 hours post dose | 40.40 [21.5 to 61.0] | 35.30 [22.8 to 51.7]
  16 hours post dose | 27.30 [16.4 to 41.6] | 26.20 [12.9 to 39.5]
  24 hours post dose | 24.50 [16.9 to 30.9] | 25.50 [12.0 to 39.3]
  48 hours post dose | 15.40 [7.86 to 22.1] | 16.20 [8.36 to 27.1]
  72 hours post dose | 12.55 [7.28 to 18.8] | 12.60 [7.50 to 27.7]
  120 hours post dose | 10.55 [4.78 to 16.3] | 11.60 [5.85 to 21.0]
  168 hours post dose | 9.120 [3.75 to 13.2] | 9.930 [4.83 to 14.9]
  216 hours post dose | 7.555 [4.10 to 14.0] | 8.150 [3.32 to 17.9]
  264 hours post dose | 7.575 [3.25 to 12.0] | 7.270 [2.75 to 13.5]
  312 hours post dose | 6.445 [2.58 to 12.7] | 6.920 [2.85 to 14.3]
  384 hours post dose | 5.180 [2.18 to 10.4] | 5.600 [1.83 to 12.7]
  456 hours post dose | 4.300 [1.65 to 8.75] | 4.330 [1.65 to 9.13]
  528 hours post dose | 3.560 [1.39 to 8.14] | 4.160 [1.03 to 10.9]

26. Secondary Outcome: Plasma Endoxifen (Metabolite) Concentration Versus Time Summary: Tamoxifen Alone and When Coadministered With DVS SR
Description: Summary statistics were to be calculated by setting concentration values below the lower limit of quantification (LLQ = 0.100 ng/mL) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) = 0.
Time Frame: as for outcome 25
Population: PK concentration analysis population. N=number of participants contributing to the median. Period 2 / Day 1 = Day 1 of Tamoxifen dosing (Period 2 / Day 7) within the DVS SR, Tamoxifen coadministration dosing period.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
ng/mL
  0 hour | NA [NA to NA] — No observations above the lower limit of quantification. | 0.2900 [0.000 to 0.799]
  0.5 hour post dose | NA [NA to NA] — No observations above the lower limit of quantification. | 0.3370 [0.000 to 0.792]
  1 hour post dose | NA [NA to NA] — No observations above the lower limit of quantification. | 0.3430 [0.000 to 1.03]
  2 hours post dose | 0.0000 [0.000 to 0.126] | 0.4100 [0.102 to 1.15]
  3 hours post dose | 0.0000 [0.000 to 0.275] | 0.5020 [0.000 to 1.14]
  4 hours post dose | 0.1760 [0.000 to 0.590] | 0.6350 [0.119 to 1.26]
  6 hours post dose | 0.2485 [0.000 to 0.516] | 0.5870 [0.000 to 1.00]
  8 hours post dose | 0.2895 [0.102 to 0.624] | 0.7310 [0.149 to 1.39]
  12 hours post dose | 0.4470 [0.116 to 0.884] | 0.7310 [0.146 to 1.39]
  16 hours post dose | 0.4330 [0.111 to 0.818] | 0.7130 [0.120 to 1.46]
  24 hours post dose | 0.6215 [0.162 to 1.05] | 0.9900 [0.203 to 1.47]
  48 hours post dose | 0.9065 [0.150 to 1.40] | 1.180 [0.270 to 2.12]
  72 hours post dose | 0.9740 [0.178 to 1.54] | 1.180 [0.208 to 1.83]
  120 hours post dose | 1.095 [0.135 to 1.89] | 1.240 [0.287 to 2.13]
  168 hours post dose | 1.120 [0.128 to 1.97] | 1.140 [0.169 to 2.23]
  216 hours post dose | 1.120 [0.149 to 1.78] | 1.080 [0.193 to 1.80]
  264 hours post dose | 1.145 [0.166 to 1.57] | 1.160 [0.168 to 1.94]
  312 hours post dose | 1.035 [0.148 to 1.69] | 0.9760 [0.157 to 1.86]
  384 hours post dose | 0.8560 [0.169 to 1.50] | 0.9470 [0.121 to 1.61]
  456 hours post dose | 0.7060 [0.104 to 1.51] | 0.9150 [0.119 to 1.37]
  528 hours post dose | 0.6210 [0.000 to 1.23] | 0.7040 [0.000 to 1.47]

27. Secondary Outcome: Plasma N-desmethyl-tamoxifen (Metabolite) Concentration Versus Time Summary: Tamoxifen Alone and When Coadministered With DVS SR
Description: as for outcome 25
Time Frame: as for outcome 25
Population: as for outcome 26
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
ng/mL
  0 hour | NA [NA to NA] — No observations above the lower limit of quantification. | 3.600 [1.22 to 8.84]
  0.5 hour post dose | 0.0000 [0.000 to 0.465] | 4.120 [1.97 to 11.2]
  1 hour post dose | 0.8050 [0.000 to 3.34] | 5.650 [2.64 to 12.4]
  2 hours post dose | 4.210 [0.310 to 9.46] | 9.770 [4.51 to 16.7]
  3 hours post dose | 9.440 [1.03 to 20.2] | 14.80 [6.30 to 26.4]
  4 hours post dose | 12.55 [2.67 to 20.7] | 18.70 [9.09 to 29.9]
  6 hours post dose | 14.10 [7.61 to 23.3] | 19.30 [11.8 to 26.1]
  8 hours post dose | 14.90 [9.97 to 23.5] | 20.40 [14.3 to 30.3]
  12 hours post dose | 16.10 [10.8 to 26.8] | 19.00 [11.1 to 25.7]
  16 hours post dose | 14.55 [9.14 to 20.1] | 18.40 [11.6 to 35.1]
  24 hours post dose | 16.90 [8.64 to 23.3] | 21.90 [12.7 to 32.4]
  48 hours post dose | 16.45 [9.49 to 23.3] | 24.00 [13.3 to 34.9]
  72 hours post dose | 16.45 [8.01 to 21.8] | 19.80 [13.9 to 31.5]
  120 hours post dose | 15.10 [8.26 to 22.9] | 19.80 [15.0 to 31.4]
  168 hours post dose | 14.40 [8.04 to 26.1] | 16.80 [12.7 to 26.3]
  216 hours post dose | 13.50 [7.75 to 19.6] | 15.60 [8.60 to 24.3]
  264 hours post dose | 12.65 [8.13 to 17.6] | 15.40 [5.80 to 22.5]
  312 hours post dose | 11.40 [6.99 to 18.0] | 14.40 [8.39 to 20.6]
  384 hours post dose | 10.15 [6.46 to 15.5] | 13.10 [6.86 to 19.7]
  456 hours post dose | 8.730 [5.35 to 14.2] | 10.50 [3.24 to 16.3]
  528 hours post dose | 8.730 [4.69 to 13.0] | 10.40 [4.36 to 21.7]

28. Secondary Outcome: Plasma 4-hydroxy-tamoxifen (Metabolite) Concentration Versus Time Summary: Tamoxifen Alone and When Coadministered With DVS SR
Description: as for outcome 26
Time Frame: as for outcome 25
Population: as for outcome 26
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Tamoxifen 40 mg (Period 1) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Number analyzed (Participants) | 30 | 29
ng/mL
  0 hour | NA [NA to NA] — No observations above the lower limit of quantification. | 0.0000 [0.000 to 0.130]
  0.5 hour post dose | NA [NA to NA] — No observations above the lower limit of quantification. | 0.0000 [0.000 to 0.171]
  1 hour post dose | NA [NA to NA] — No observations above the lower limit of quantification. | 0.0000 [0.000 to 0.321]
  2 hours post dose | 0.2060 [0.000 to 0.431] | 0.2030 [0.000 to 0.633]
  3 hours post dose | 0.4335 [0.000 to 0.811] | 0.3960 [0.136 to 1.00]
  4 hours post dose | 0.5900 [0.101 to 1.03] | 0.6420 [0.232 to 1.13]
  6 hours post dose | 0.6145 [0.346 to 0.889] | 0.7060 [0.340 to 0.985]
  8 hours post dose | 0.6290 [0.307 to 0.985] | 0.7100 [0.408 to 1.06]
  12 hours post dose | 0.5910 [0.312 to 0.966] | 0.5860 [0.354 to 1.07]
  16 hours post dose | 0.4920 [0.322 to 0.887] | 0.5640 [0.308 to 0.947]
  24 hours post dose | 0.5395 [0.329 to 0.930] | 0.5780 [0.300 to 1.02]
  48 hours post dose | 0.4925 [0.233 to 0.931] | 0.4910 [0.235 to 1.12]
  72 hours post dose | 0.3795 [0.174 to 0.717] | 0.4010 [0.200 to 0.903]
  120 hours post dose | 0.2845 [0.102 to 0.627] | 0.2920 [0.171 to 0.745]
  168 hours post dose | 0.2180 [0.000 to 0.525] | 0.2270 [0.107 to 0.548]
  216 hours post dose | 0.1840 [0.000 to 0.435] | 0.1870 [0.000 to 0.423]
  264 hours post dose | 0.1590 [0.000 to 0.361] | 0.1600 [0.000 to 0.367]
  312 hours post dose | 0.1315 [0.000 to 0.338] | 0.1380 [0.000 to 0.323]
  384 hours post dose | 0.1125 [0.000 to 0.280] | 0.1180 [0.000 to 0.286]
  456 hours post dose | 0.0000 [0.000 to 0.283] | 0.0000 [0.000 to 0.208]
  528 hours post dose | 0.0000 [0.000 to 0.230] | 0.0000 [0.000 to 0.296]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 36 (follow-up telephone visit)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. Participants are counted for each treatment sequence.
Groups:
- Tamoxifen 40 mg (Period 1): Tamoxifen 40 mg as a single oral dose on Period 1 / Day 1.
- DVS SR 100 mg (Period 2): DVS SR 100 mg as a single oral daily dose Period 2 / Day 1 through Day 6 (steady state) and Day 7 through Day 28.
- Tamoxifen 40 mg + DVS SR 100 mg (Period 2): Tamoxifen 40 mg as a single oral dose coadministered with DVS SR 100 mg as a single oral dose on Period 2 / Day 7.
Arm/Group | Tamoxifen 40 mg (Period 1) | DVS SR 100 mg (Period 2) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2)
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 11/30 | 17/29 | 24/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tamoxifen 40 mg (Period 1) (N=30) | DVS SR 100 mg (Period 2) (N=29) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2) (N=29)
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tamoxifen 40 mg (Period 1) (N=30) | DVS SR 100 mg (Period 2) (N=29) | Tamoxifen 40 mg + DVS SR 100 mg (Period 2) (N=29)
Palpitations (Cardiac disorders) | 0 | 0 | 7
Eye swelling (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 4
Vaginitis bacterial (Infections and infestations) | 0 | 1 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 3
Headache (Nervous system disorders) | 1 | 1 | 9
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 2 | 8
Nightmare (Psychiatric disorders) | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.